CLINICAL TRIAL: NCT04669522
Title: How do Psychological Factors Interact With the Oncological Outcomes of Women With Triple-negative Breast Cancer?
Brief Title: Psychological Factors and Oncological Outcomes of Triple-negative Breast Cancer
Acronym: PSY-ONC TNBC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pius-Hospital Oldenburg (Other)
Collaborators: University of Oldenburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. med. Rudy Leon De Wilde, Clinic Director, Pius-Hospital Oldenburg
Other Study IDs: PHDW-006
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Psychooncology
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been established that chronic stress can take a toll on one's health. Furthermore, when an someone falls ill, it is believed that the way that they handle stress and/or adversity can positively or negatively impact the course of their disease. Against the background of these findings, this study aims to explore how (1) cumulative lifetime stress exposure, (2) coping response, (3) perceived social support, and (4) and overall psychological well-being may relate to the oncological outcomes of women diagnosed with triple negative breast cancer (TNBC).

Patients treated for TNBC between 01.01.2015-31.12.2019 at the University Clinic for Gynecology at Pius-Hospital Oldenburg will be asked to complete four questionnaires corresponding to the abovementioned psychological aspects. The results of these questionnaires will be analyzed together with the clinical patient data and tumor characteristics (such as type, size, etc.) to explore whether there is a tendency between one or more of the above-mentioned psychosocial aspects and the course of the disease (e.g. a disease recurrence within one year after the initial diagnosis (yes / no), the duration of the disease-free or progression-free period).

As there is an existing body of evidence supporting a relationship between stress and the immune system, we expect to see the poorest oncological outcomes in patients who 1) have faced more stressful/adverse life events, 2) those who present inadequate/inappropriate coping skills, 3) report less social support, and 4) poorer overall psychological well-being.

If a potential connection between psychosocial factors and the course of the TNBC is identified, further disease specific, it will aid in the development of disease-specific, health-promoting measures to better support this particular patient group. This is of great importance, as TNBC is generally associated with clinically aggressive behavior and a worse prognosis compared to other breast cancer subtypes.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) is a highly heterogeneous subtype, which exhibits aggressive clinical behavior and generally carries a poor prognosis. As it lacks hormone receptors expression (estrogen and progesterone receptors) and amplification of the Human epidermal growth factor receptor 2 (HER2), targeted therapies are lacking. Thus, the identification of any modifiable factors which may influence the course of the disease is critical both in improving the quality of care and the patient's quality of life. In addition to lifestyle factors, such as diet and exercise habits, psychological factors, such as cumulative lifetime stress, coping response, perceived social support, and overall psychological well-being may also influence cancer progression.

While it is known that stress can directly upregulate certain immune mechanisms, it is suspected that a patient's coping response, perceived social support, and general psychological well-being may have an indirect influence on cancer progression via altered health-related behaviors. For example, during stressful periods, alcohol consumption may rise, sleep quality may be diminished, nutritional needs may not be properly met, and exercise may be avoided. As a group, TNBC patients face additional challenges not experienced by other BC patients. Due to the disease's poor prognosis, its relatively new status as a BC subtype (first mention in 2005), and the lack of targeted treatments; patients may experience an increased stress-response following their diagnosis. For instance, it is known that an event induces a stress response when it involves novelty and unpredictability, a lack of sense of control, and threats to the sense of self; elements that are clearly emphasized in TNBC.

To promote the development of psycho oncological strategies tailored towards women in this particular patient group, this study aims to explore any trends which might be indicative of an interaction between psychological aspects and the oncological outcomes of patients treated for TNBC between 01.01.2015-31.12.2019, at Pius Hospital, in Oldenburg, Germany. Because we intend to evaluate a retrospective cohort of patients, the psychological instruments were chosen and slightly adapted to target past events (stress across life span and social support) and stable traits (psychological well-being, coping).

As there is an existing body of evidence supporting the relationship between stress and the immune system, we expect to see the poorest oncological outcomes in patients who 1) have had more adverse life events, and 2) those who present inadequate/inappropriate coping skills. Additionally, we intend to explore if other psychological variables mentioned in the literature, including perceived social support and psychological well-being, are also related to the oncological outcomes in our cohort of patients.

This study combines prospective and retrospective approaches since the psychosociological data is to be collected prospectively from a single retrospective cohort of patients. Patients could not be randomized into groups, due to the retrospective nature of the study. Considering that all data derived from this study will be numerical, this will be a quantitative analysis. This research is comparative since the patients' clinical outcomes will be analyzed in terms of psychological measures. Lastly, the present study is exploratory as it aims to shed light on the interplay between psychological and clinical aspects in TNBC, as psycho-oncological studies are lacking for this BC subtype.

A list of patient names will be obtained from the hospital's Tumor Documentation Office. Next, patient electronic medical records will be accessed through Pius-Hospital's Orbis Database program according to the name and date of birth of each patient. Demographic and clinical variables of interest will be collected from the clinical charts and recorded on the patient case report form (CRF).

The psychological aspects of interest will be assessed through self-reported questionnaires. (1 computer-based and 3 paper-based questionnaires). Patients will fill out the surveys in a proper setting where privacy will be assured. Questionnaires will not include information which could be directly used to identify participants (i.e. name, DOB), but will instead contain a code which will allow the psychological data to be combined with the respective participant's demographic and clinical variables for the subsequent statistical analysis. After completion, participant's information (pseudonymized) will be transferred to the CRF, and subsequently case data will be transferred to SPSS (software version 26.0) for further statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of TNBC, with the ability to speak and understand German, who can give informed consent, and who were treated in the University Hospital for Gynecology, Pius-Hospital Oldenburg, between 01.01.2015-31.12.2019

Exclusion Criteria:

* 1) any woman with an unconfirmed TNBC diagnosis, 2) woman whose medical records are lacking clinical and/or pathological variables of interest, 3) patients with current or previous mood disorder, psychosis, anxiety disorder, psychosis, anxiety disorder, or substance abuse disorder according to the DSM V, Diagnostic and Statistical Manual of Mental Disorders, and 5) all women who currently make use of psychotropic agents or psychiatric drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective cohort will be composed of a minimum of 50 patients diagnosed with TNBC and treated in the University Hospital for Gynecology, Pius-Hospital Oldenburg, between 01.01.2015-31.12.2019.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall Severity Score (OSS) | 1 day
  Cumulative lifetime stress will be quantified as a score (Overall Severity Score; OSS) derived from the Stress and Adversity Inventory (STRAIN) questionnaire (Slavich and Shields, 2018).

SECONDARY OUTCOMES:
Hazard ratio associated with OSS | 1 day